CLINICAL TRIAL: NCT04337073
Title: The Effect of Propofol on Dexamethasone-induced Perineal Pruritus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Ma Hong, Affiliated hospital of Yangzhou university, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MHong
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Pruritus
Keywords: propofol; Dexamethasone; pruritus
MeSH Terms: conditions — Pruritus | interventions — Propofol; Saline Solution

STUDY DESIGN:
Intervention Model Description: propofol (P) group and normal saline (N) group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal saline (N) group (Placebo Comparator): Before anesthesia induction, N group received corresponding intravenous normal saline of the same volume.
  Interventions: Drug: normal saline
- propofol (P) group (Active Comparator): Before anesthesia induction, P group received intravenous injection of 0.3mg/kg propofol
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Before anesthesia induction, M group received intravenous injection of 0.3mg/kg Propofol, while N group received corresponding intravenous normal saline of the same volume. After 1 min, both groups received intravenous injection of dexamethasone sodium phosphate injection of 10mg.
  Arms: propofol (P) group
Drug: normal saline — Before anesthesia induction, M group received intravenous injection of 0.3mg/kg Propofol, while N group received corresponding intravenous normal saline of the same volume. After 1 min, both groups received intravenous injection of dexamethasone sodium phosphate injection of 10mg.
  Arms: normal saline (N) group

SUMMARY:
patients may appear serious perineal itching, after injection of dexamethasone sodium phosphate injection its incidence is about 25% ~ 100%, and the incidence of the discomfort in females was much higher than that of the maleTo investigate the effect of propofol pretreatment on perineal pruritus induced by dexamethasone sodium phosphate injection and explore the possible machanisms.

DETAILED DESCRIPTION:
40 patients scheduled for selective surgery,aged 18-65years,ASA physical status I~II,BMI 18~30kg/m2 were selected in this study.The patients were equally randomized into two groups: propofol (P) group and normal saline (N) group, 20 cases in each group. Before anesthesia induction, M group received intravenous injection of 0.3mg/kg propofol , while N group received corresponding intravenous normal saline of the same volume. After 1 min, both groups received intravenous injection of dexamethasone sodium phosphate injection of 10mg. The anesthesiologist assessed perineal irritation in both groups and recorded Ramsay scores,the number of cases, visual analogue scale(VAS) scores ,duration of itching and observed the occurrence of adverse reactions such as dizziness, hypotension and respiratory depression in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Elective female surgery patients, ages 18 to 65 years old, ASA Ⅰ or Ⅱ level, body mass index (BMI) of 18 ~ 30 kg/m2.

Exclusion Criteria:

* diabetes mellitus, paresthesia, allergy to narcotic drugs, routine preoperative use of narcotic analgesics, long-term use of hormones, drug and alcohol abuse, communication disorders in psychiatric disorders, pregnancy or lactation, and patients with severe systemic diseases and unwilling to undergo the trial.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 40 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
visual analogue scale(VAS) scores | in 3min
  VAS score was used to grade the degree of perineal itching: VAS 0 was no discomfort, 1-3 was mild, 4-6 was moderate, and 7-10 was severe

SECONDARY OUTCOMES:
the occurrence of adverse reactions | in 3min
  the occurrence of adverse reactions such as dizziness, hypotension and respiratory depression in the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated hospital of yangzhou university, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No